CLINICAL TRIAL: NCT06060340
Title: Clinical and Radiographic Outcomes of Class II Furcation Defects Management Using Propolis: A Case Series
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Said Abd-El Azeem Allam, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERIO 3-3-2
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Furcation Defects
MeSH Terms: conditions — Furcation Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- class II furcation defects (Experimental): Inclusion criteria:
  1. Lower molars with class II furcation defects.
  2. Full mouth plaque score (FMPS )<20% at baseline.
  3. Full mouth bleeding score (FMBS )<10% at baseline.
  4. Systemically healthy.
  5. Cooperative patients.
  Exclusion criteria:
  1. Smokers.
  2. Pregnancy and lactation.
  3. Stage 4 Grade C periodontitis.
  Interventions: Drug: class II furcation defects management using propolis

INTERVENTIONS:
Drug: class II furcation defects management using propolis — A full thickness flap will be elevated using muco-periosteal elevator to gain full access to the furcation defect. Then granulomatous tissue will be debrided from the osseous defect and the root surfaces will be carefully scaled and root planed by ultrasonic and hand instruments.
  The diagnosis of the class II furcation defect was then confirmed using a Naber's probe.
  Propolis preparation:
  Pure propolis will then be mixed with saline to give a proper mix/consistency and applied to completely fill the furcation defect.

SUMMARY:
Furcation involvement represents a challenge for treatment to many periodontists due to many factors including access, morphology, and variations of anatomical features of the furcation area. Furcation involvement treatment includes non-surgical periodontal therapy, resective surgery and regenerative surgery, regenerative therapy utilizing different graft materials and membranes is of high cost and research for new materials that can be cost-effective and available for all patients is continuing, propolis have been shown to be cost-effective therapy for bone and wound healing.

DETAILED DESCRIPTION:
Propolis is a natural resinous product of the bee workers collected from trees to use it to stick their hives and form a coat to protect their hives from all sources of bacteria and invasions. Propolis is composed of more than 300 compounds, the most important of them are flavonoids like CAPE (caffeic acid phenyl ester). Propolis have shown anti-inflammatory, anti-oxidant, anti-bacterial, anti-fungal, anti-viral and more importantly regenerative effect and bone formation capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Lower molars with class II furcation defects.
  2. Full mouth plaque score (FMPS )<20% at baseline.
  3. Full mouth bleeding score (FMBS )<10% at baseline.
  4. Systemically healthy.
  5. Cooperative patients.

Exclusion Criteria:

* Exclusion criteria:

  1. Smokers.
  2. Pregnancy and lactation.
  3. Stage 4 Grade C periodontitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Horizontal and Vertical Clinical Attachment Level (CAL) | 6 months
  Measured from the CEJ to the bottom of the gingival sulcus using Naber's periodontal probe.
  Measured from the CEJ to the bottom of the gingival sulcus using William's periodontal probe.

SECONDARY OUTCOMES:
Radiographic Defect Fill | 6 months
  The depth of Furcation defect will be measured from the Furcation to the base of the defect at baseline and after six months to detect the amount of bone fill. Individually customized bite blocks will be created for the patients using alginate impression material and acrylic resin. Parallel-angle technique will be used to obtain standardized radiographs
Probing Depth (PD) | 6 months
  Measured from the gingival margin to the bottom of the gingival sulcus using William's periodontal probe with the probe inserted parallel to the long axis of the tooth
Bleeding on Probing (BOP) | 6 months
  BOP score will be assessed as the number of bleeding sites (dichotomous yes/no evaluation) when stimulated by a standardized periodontal probe with a controlled (∼25 g) force to the bottom of the sulcus at six sites (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, disto-lingual) on all present teeth
Plaque Index (PI) | 6 months
  PI will be assessed using a standardized periodontal probe to agitate the gingival margin and assessing the presence or absence of plaque at the margin. This will be recorded at 4 sites per tooth on all teeth
Gingival Recession | 6 months
  Measured from the cementoenamel junction to the gingival margin using a William's graduated periodontal probe. The probe will be inserted into the sulcus gently parallel to the long axis of the tooth

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, El-Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
one arm (10 participents)
  Inclusion criteria:
  1. Lower molars with class II furcation defects.
  2. Full mouth plaque score (FMPS )<20% at baseline.
  3. Full mouth bleeding score (FMBS )<10% at baseline.
  4. Systemically healthy.
  5. Cooperative patients.
  Exclusion criteria:
  1. Smokers.
  2. Pregnancy and lactation.
  3. Stage 4 Grade C periodontitis.